**Document Type:** Informed Consent Form

Official Title: Barriers and Facilitators to Following the Dietary Guidelines for Vegetable Intake: Follow-up

of an Intervention to Increase Vegetable Consumption

NCT Number: NCT03607526

**IRB Approval Date:** 05/08/2019

# THE UNIVERSITY OF NORTH DAKOTA CONSENT TO PARTICIPATE IN RESEARCH

TITLE: Barriers and Facilitators to Vegetable Intake

**PROJECT DIRECTOR:** Angela De Leon, PhD

PHONE # 701-795-8148

**DEPARTMENT:** ARS-USDA Human Nutrition Research Center

#### STATEMENT OF RESEARCH

A person who joins this study must give his or her informed consent. This consent must be based on an understanding of the nature and risks of the research. This document provides information that is important for this understanding. Only people who want to take part in a research study may do so. Please take your time in making your decision as to whether to participate. If you have questions at any time, please ask.

#### WHAT IS THE PURPOSE OF THIS STUDY?

You are invited to be part of this study because you were part of another study here at the Grand Forks Human Nutrition Research Center (GFHNRC) and gave us permission to contact you for a future study.

The purpose of this study is to find out why people do or do not eat vegetables. You will meet in a group of 6-9 people. There will be 8 groups.

## **HOW MANY PEOPLE WILL PARTICIPATE?**

A total of 48-72 people will take part in this study at the USDA GFHNRC.

## HOW LONG WILL I BE IN THIS STUDY?

Your part of the study will take about 2 hours.

#### WHAT WILL HAPPEN DURING THIS STUDY?

At the group meeting you will be asked a question about things that make it hard or easy to eat vegetables. Without using names, we will take notes to help us recall the main points of each discussion. You will not be recorded on tape or video.

| Approval Date: | MAY | 8 | 2 | 2019 |
|--------------------------------|-----|---|---|------|
| Expiration Date: _ | MAY | 7 | 1 | 2020 |
| University of North Dakota IRB | | | | |

| Date: |
|-------------------|
| Subject Initials: |

## WHAT ARE THE RISKS OF THE STUDY?

The risk for being in this study is very small. You may feel nervous about speaking in front of people and having people hear your ideas.

#### WHAT ARE THE BENEFITS OF THIS STUDY?

You will not benefit from being in this study. However, other people might benefit from this study because we will learn more about why people do or do not eat vegetables.

## WILL IT COST ME ANYTHING TO BE IN THIS STUDY?

We do not withhold taxes from any monies you receive. Any questions you have related to taxes will need to be directed to your personal accountant or the Internal Revenue Service.

## WILL I BE PAID FOR PARTICIPATING?

You will be paid \$40 for being in the study.

#### WHO IS FUNDING THE STUDY?

The United States Department of Agriculture is funding this research study. No one on the research team will receive a direct payment or an increase in salary for conducting this study.

## **CONFIDENTIALITY**

The records of this study will be kept private to the extent permitted by law. In any report about this study that might be published, the study results will be in a summarized manner and you will not be identified. None of the study results will have any names attached. The consent and the check information will be kept in a locked file at the Grand Forks Human Nutrition Research Center.

Your records may be reviewed in order to meet federal or state regulations. Reviewers may include the US Department of Agriculture as specified in the USDA/ARS Privacy Act System of Records, the UND Research Development and Compliance office, and the University of North Dakota Institutional Review Board.

#### IS THIS STUDY VOLUNTARY?

Your participation is voluntary. You may choose not to join or you may stop at any time without penalty or loss of benefits that you are otherwise allowed. Your decision whether or not to participate will not affect your current or future relations with the GFHNRC or the University of North Dakota.

| Approval Date: | MAY | 8 | 2019 |
|--------------------------------|-----|---|------|
| Expiration Date: | MAY | 7 | 2020 |
| University of North Dakota IRB | | | |

| Date: |
|-------------------|
| Subject Initials: |

# **CONTACTS AND QUESTIONS**

The scientist conducting this study is Angela De Leon. You may ask any questions you have now. If you later have questions, concerns, or complaints about the research please contact Dr. De Leon at <a href="mailto:angela.deleon@ars.usda.gov">angela.deleon@ars.usda.gov</a> or by phone at 701-795-8148.

If you have questions regarding your rights as a research subject, you may contact The University of North Dakota Institutional Review Board at (701) 777-4279 or <a href="mailto:UND.irb@research.UND.edu">UND.irb@research.UND.edu</a>.

- You may also call this number about any problems, complaints, or concerns you have about this research study.
- You may also call this number if you cannot reach research staff, or you wish to talk with someone who is independent of the research team.
- General information about being a research subject can be found by clicking "Information for Research Participants" on the web site: <a href="http://und.edu/research/resources/human-subjects/research-participants.cfm">http://und.edu/research/resources/human-subjects/research-participants.cfm</a>

## **CONSENT**

Informed consent is required of all persons who participate in research studies. Your signature indicates that this research study has been explained to you, that your questions have been answered, and that you agree to take part in this study. You will receive a copy of this form.

| Subjects Name: | |
|---|---|
| Signature of Subject | Date |
| I have discussed the above points with the subject legally authorized representative. | or, where appropriate, with the subject's |
| <br>Signature of Person Who Obtained Consent | Date |

| Approval Date: | MAY | 8 | 2019 |
|--------------------------------|-----|---|------|
| Expiration Date: _ | MAY | 7 | 2020 |
| University of North Dakota IRB | | | |

| Date: |
|-------------------|
| Subject Initials: |